CLINICAL TRIAL: NCT01716052
Title: Women's Mammography Study Attempting to Improve the Comfort During Screening Mammography CTRC#11-45
Brief Title: Women's Mammography Study To Improve Comfort During Mammography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Kenneth A. Kist, (Other)
Responsible Party: Sponsor-Investigator, Kenneth A. Kist,, Principal Investigator, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTRC 11-45; HSC20120142H (Other: UTHSCSA IRB)
Record Dates: First submitted 2012-10-18; First posted 2012-10-29 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Pain
Keywords: Mammogram; Ibuprofen; Pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen (Active Comparator): Pfizer 200 mg caplets (Advil)
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator): Lactulose
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Lactulose
  Arms: Placebo
Drug: Ibuprofen
  Arms: Ibuprofen

SUMMARY:
The purpose of this study is to determine in a randomized trial whether it is possible to decrease the discomfort of mammography by using the analgesic ibuprofen, or by using a scripted, supportive text informing patients about mammography.

DETAILED DESCRIPTION:
This study is designed to evaluate two methods of reducing pain and discomfort caused by mammography, one of the barriers to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must have signed the informed consent.
* Must either be getting her first mammogram or based on prior experience be expecting level 4 or 5 pain

Exclusion Criteria:

* May not have taken ibuprofen or other pain medication within the last 12 hours.
* Must not have a contraindication for taking ibuprofen e.g:
* No history of allergic reactions to ibuprofen or aspirin
* No recent history with the last year of bleeding from GI tract
* Not pregnant or suspected of being pregnant

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kist, MD, Principal Investigator — University of Texas
Locations (1):
- Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: When the woman signs in at the breast imaging clinic desk (on the 5th floor of the Zeller Building at the CTRC), she will be asked if she would speak with the study nurse about this study.
Groups:
- Ibuprofen: Pfizer 200 mg caplets (Advil)
  Ibuprofen
Period: Overall Study
Arm/Group | Ibuprofen | Placebo
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Withdrawal of funding | 1 | 1

BASELINE CHARACTERISTICS:
Population: Two sided significance level of 0.05 and a statistical power of 0.90 with 187 patients in both the placebo and the ibuprofen group..
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Measure of Discomfort of Mammography
Description: The primary outcome measure will be the response to questions on a questionnaire.
Time Frame: 3 years
Population: No data was collected or analyzed for the outcome measure because the study was terminated.
Arm/Group | Ibuprofen | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Total number of participants at risk is "0" since adverse events were not collected/assessed.
Arm/Group | Ibuprofen | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No